CLINICAL TRIAL: NCT00514033
Title: Open, Multicentric, PMS Study to Monitor Safety and Reactogenicity of GlaxoSmithKline Biologicals' Poliomyelitis Vaccine (Inactivated)-Poliorix, Administered in Korean Children as a Primary Vaccination in Healthy Subjects Aged 2 to 6 Months or as a Booster Vaccination in Subjects Aged 4 to 6 Years
Brief Title: A Post-marketing Safety Study of GSK Bio IPV Vaccine (PoliorixTM) in Korean Children
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 108344
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Poliomyelitis
MeSH Terms: conditions — Poliomyelitis | interventions — Poliovirus Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Group A: PoliorixTM will be administered according to a 3-dose schedule at 2, 4, 6 months for primary vaccination followed by a booster dose between 4 to 6 years. For the primary vaccination course, 1 to 3 doses of the vaccine will be given depending on previous vaccination history with poliomyelitis vaccine.
  Interventions: Biological: Poliomyelitis vaccine (inactivated) -PoliorixTM

INTERVENTIONS:
Biological: Poliomyelitis vaccine (inactivated) -PoliorixTM — Deep intramuscular injections for the primary vaccination and booster vaccination.

SUMMARY:
Following licensing of PoliorixTM in Korea, this study will collect safety data about the routine use of this vaccine in 600 children according to the regulations of Korean Food and Drugs Administration (KFDA).

DETAILED DESCRIPTION:
An open, multicentric, post-marketing surveillance study to monitor the safety and reactogenicity of GlaxoSmithKline Biologicals. Poliomyelitis vaccine (inactivated) -PoliorixTM., administered in Korean children as a primary vaccination in healthy subjects aged two to six months or as a booster vaccination in subjects aged four to six years.

ELIGIBILITY:
Inclusion Criteria:

* A healthy male or female child between two and six months of age (primary vaccination) or between four and six years of age (booster vaccination) at the time of vaccination.
* Subjects for whom the investigator believes that their parents/guardians can and will comply with the requirements of the protocol (e.g. completion of the diary cards)
* Written informed consent obtained from the parent/ guardian of the subject

Exclusion Criteria:

* At the time of study entry, the contraindications and precautions of use indicated in the Korean Label should be checked and the subject must not be included in the study if there is any contraindication or risk

Ages: 2 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Korean children between two and six months of age (primary vaccination) or between four and six years of age (booster vaccination) at the time of vaccination.
Sampling Method: Probability Sample
Enrollment: 349 (Actual)
Dates: Start 2007-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of unsolicited adverse events. | During 7 days (Day 0 - 6) following vaccination.
Occurrence of serious adverse events (SAEs). | During the entire study period.

SECONDARY OUTCOMES:
Occurrence of solicited local and general adverse events. | During 7 days (Day 0 to 6) after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Seoul, South Korea